CLINICAL TRIAL: NCT03791073
Title: Discovery of New Biomarkers in Pancreatic Cancer Using Novel Nondestructive OMICS Methodology
Brief Title: New Biomarkers in Pancreatic Cancer Using EXPEL Concept
Acronym: PANEXPEL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: IRCM U1194 INSERM, Tumor Microenvironment and Resistance to Treatment Lab (Unknown); IRCM U1194 INSERM, Cancer Bioinformatics and Systems Biology's team (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0437
Record Dates: First submitted 2018-12-13; First posted 2019-01-02 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Oncology
Keywords: Biomarker discovery; Pancreatic adenocarcinoma; Bioinformatics; pancreatic cancer; microenvironment; proteomics; transcriptomics; metabolomics; diagnosis; Prognosis
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cytolyt Samples:
  Liquid conservation samples from patients who underwent endoscopic ultrasound with fine needle aspiration/biopsy for suspicious pancreatic mass at the CHU de Montpellier were conserved at +4°c.
  Cytolyt samples do not contain any cell or tissue from patient, this liquid is systematically trashed in current practice. No genetics analysis will be performed from these particular samples in the present study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators recently engineered a novel biomarker discovery approach that is non-destructive and fully compatible with OMICS profiling as well as routine clinical procedures (5). The latter approach - termed EXPEL - mines the interstitial tissue fluid that is the richest source of soluble, undiluted and uncontaminated biomarkers. The method notably gives access to proteins, metabolites, RNA, DNA and exosomes, thus enabling holistic biomarker discovery. Owing to its non-destructive nature, EXPEL provides for the first time both clinicians and researchers with the opportunity to analyze identical material.

The investigators hypothesize that the conservation liquid used to collect cells and biopsy after endoscopic ultrasound for pancreatic biopsy could contain the tissue secretome and permit a comprehensive OMICS analysis of PDAC (all stages confounded) by using a "modified EXPEL" procedure. These are ideal conditions for EXPEL approach that will additionally to finding novel biomarkers also shed light on complex network of cancer cell-stroma interactions.

DETAILED DESCRIPTION:
Biomarkers that are readily detectable in fluid biopsies are of outmost importance for diagnosis and prediction of therapeutic response in all cancer patients. Pancreatic ductal adenocarcinoma (PDAC) is an example of a deadly malignancy that is diagnosed very late due to lack of sensitive and reliable markers [1]. The incidence and mortality of PDAC will double in the next 15 years, which is unprecedented among all cancer types [2]. Secondary cancer prevention through early diagnosis of PDAC will therefore be an essential preparedness asset for facing the immense healthcare burden.

Discovery of diagnostic biomarkers depends essentially on the availability of patient material ideally collected at different time points during the disease progression (e.g. early lesion, before treatment and after recurrence). Unfortunately, it is very difficult to access fresh biopsies from pre-malignant lesions for research purposes. These are needed in their entirety for histo-pathological evaluation and diagnosis. The ability to use liquid biopsies (e.g. serum, urine, saliva) brought the promise to circumvent this problem, opening access to many different biomolecules such as circulating DNA and proteins. However, upon their release from the tumor, these molecules are diluted up to several billion-fold in blood with molecular species originating from healthy tissues [3-4]. This hampers de novo discovery of biomarkers for diagnosing and understanding the disease.

To circumvent these limitations, the investigators recently engineered a novel biomarker discovery approach that is non-destructive and fully compatible with OMICS profiling as well as routine clinical procedures (5). The latter approach - termed EXPEL - mines the interstitial tissue fluid that is the richest source of soluble, undiluted and uncontaminated biomarkers. The method notably gives access to proteins, metabolites, RNA, DNA and exosomes, thus enabling holistic biomarker discovery. Owing to its non-destructive nature, EXPEL provides for the first time both clinicians and researchers with the opportunity to analyze identical material, while having virtually no disadvantage in their respective tasks. The investigators have recently shown the ability of our methodology to find new markers in the context of precious human colorectal cancer samples. Thus, the investigators are convinced that EXPEL can be successfully applied to pancreatic cancer. In addition, knowing the important proportion of stroma in PDAC (usually 2/3 of tumor mass), the secretome of pancreatic cancer is expected to be much richer in soluble "communication factors" exchanged between cancer cells and host tissue.

In clinical practice, most of patients undergo endoscopic ultrasound with fine needle aspiration/biopsy of the pancreatic mass to confirm the diagnosis of PDAC. The needle is rinsed in a conservation liquid Cytolyt® (Methanol 30% et water 50%) and sent to the pathologists. Microbiopsy are fixed in paraffin then analyzed and liquid is cytofiltrated to keep potential tumor cells. The remnant Cytolyt® liquid is systematically trashed.

The present study is based on the hypothesis that this liquid, previously in contact with tumoral tissue, could contain the tissue secretome and permit a comprehensive OMICS analysis of PDAC (all stages confounded) by using a "modified EXPEL" procedure. These are ideal conditions for EXPEL approach that will additionally to finding novel biomarkers also shed light on complex network of cancer cell - stroma interactions.

For this purpose, the investigators aim to perform proteomic analysis on the conservation liquid (Cytolyt) in patients who underwent endoscopic ultrasound with fine needle aspiration/biopsy for suspicious pancreatic mass at the CHU de Montpellier between Jan 2018 and Jan 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pancreatic mass and suspicion of pancreatic ductal adenocarcinoma requiring endoscopic ultrasound with fine needle biopsy or surgery
* Patient ≥18 years old
* Patient naïve of any treatment of Pancreatic cancer

Exclusion Criteria:

* Patient who reject the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pancreatic mass and suspicion of pancreatic ductal adenocarcinoma requiring endoscopic ultrasound with fine needle biopsy or surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Predictive value of each protein contained in Cytolyt® for the positive diagnosis of pancreatic ductal adenocarcinoma | an average of 1 year
  Correlation with positive diagnosis of pancreatic ductal adenocarcinoma and proteins quantity in Cytolyt® samples using ROC curves (sensibility/specificity: Area Under the Curve > 0.85) and binary logistic regression method with controlling for the effects of the co-variates (such as age, disease cTNM stage, and treatment details).

SECONDARY OUTCOMES:
Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis | 1 year
  Disease-free survival (percentage of patients without recurrence) at 1 year
Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis | 1 year
  Overall survival at 1 year (percentage of patients alive)
Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis | 1 year
  Disease-free survival (DFS) (time from diagnosis to time of first radiological evidence of local, regional, or distant relapse, or death due to any cause)
Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis | 1 year
  Overall survival (OS) (time from diagnosis until death, regardless of cause)
Biomarkers that are prognostically significant on disease free or overall survival in patients with pancreatic cancer, identified using the survival analysis | 1 year
  Kaplan Meier analysis, logrank test and Cox's proportional hazards regression model to identify biomarkers that are prognostically significant (Hazard ratio (HR) and its 95% confidence interval (CI)).

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

REFERENCES:
- [Derived] Souche R, Tosato G, Riviere B, Valats JC, Debourdeau A, Flori N, Pourquier D, Fabre JM, Assenat E, Colinge J, Turtoi A. Detection of soluble biomarkers of pancreatic cancer in endoscopic ultrasound-guided fine-needle aspiration samples. Endoscopy. 2022 May;54(5):503-508. doi: 10.1055/a-1550-2503. Epub 2021 Aug 26. PMID 34448184